CLINICAL TRIAL: NCT06271005
Title: Neurological Dry Eye Study Stimulating Both Lacrimal and Vagus Nerves
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Genetic Disease Investigators (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000824
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Disease; Dry Eye
Keywords: vagus nerve; Ehlers-Danlos Syndrome; EDS; lacrimal nerves; dry eye; tear production; dysautonomia; POTS; Postural Orthostatic Tachycardia Syndrome; constipation; gastroparesis; tachycardia; NeuroTears; Mast Cell Activation Syndrome; vagus nerve stimulation; MCAS; Post-COVID; COVID; Longhaulers
MeSH Terms: conditions — Dry Eye Syndromes; Ehlers-Danlos Syndrome; Lacerations; Autonomic Nervous System Diseases; Postural Orthostatic Tachycardia Syndrome; Constipation; Gastroparesis; Tachycardia; Mast Cell Activation Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with NeuroTears (Active Comparator)
  Interventions: Dietary Supplement: NeuroTears
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NeuroTears — Over-the-counter supplement
  Arms: Treatment with NeuroTears
Dietary Supplement: Placebo — Oral placebo pill
  Arms: Placebo

SUMMARY:
This is a study on neurological dry eye disease, focusing on a patented over-the-counter supplement supporting tear production neurologically, including the lacrimal and vagus nerves.

DETAILED DESCRIPTION:
Chronic inflammation is implicated in the majority of chronic dry eyes. The parasympathetic nervous system is responsible for both basal tear secretion (the aqueous layer) by the lacrimal functional unit, and is responsible for controlling many aspects of chronic inflammation via the vagus nerve.

This study will document its effects on dry eyes, in addition to other symptoms/signs of low parasympathetic nervous system functioning using an over-the-counter supplement.

ELIGIBILITY:
Inclusion Criteria:

* Must have dry eye (OSDI score 30 and above)
* Tear break up time of less than or equal to 7 seconds
* Must be able to come for baseline tests and again at 4 weeks

Exclusion Criteria:

* Demodex
* Corneal scarring
* must not take Physostigmine (glaucoma), Pyridostigmine (Mestinon), Neostigmine (for Myasthenia Gravis); Aricept (for Alzheimer's), or ingredients to NeuroTears
* No known allergies to ingredients in NeuroTears

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | 4 weeks
  Ocular Surface Disease Index